CLINICAL TRIAL: NCT02286375
Title: Health-social Partnership Intervention Programme for Community-dwelling Older Adults: a Randomized Controlled Trial
Brief Title: Effects of Health-social Partnership Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frances Kam Yuet WONG (Other)
Responsible Party: Sponsor-Investigator, Frances Kam Yuet WONG, Professor, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSPP-01
Record Dates: First submitted 2014-10-08; First posted 2014-11-07 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Health Behavior
Keywords: health-social partnership; self-efficacy
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Interventions include providing comprehensive assessment from Omaha system, giving information regarding the self-care management, assisting and coordinating self-regulating skills and abilities, and providing social support from health-social care team to community-dwelling older adults for three months
  Interventions: Behavioral: Intervention group
- customary care group (Placebo Comparator): Customary care includes receiving community services from the community center in the district, providing monthly social call by a reserch assistant for three months
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — A structured assessment is conducted using the Omaha system. Problems will be identified in the four domains which include environment, psychosocial, physiological and health-related behavior. According to the identified problems, the nurse case manager and older adults will set contract goals and formulate an individual care plan. The nurse case manager will provide information on the basic knowledge of participants' own chronic illnesses; recognition, measurement and management of the early signs and symptoms of a deterioration or exacerbation of diseases; and the importance of health-promoting and self-care activities. A booklet will be given to them for easy reference and act as a reminder to consolidate the knowledge in case the important concepts are forgotten.

SUMMARY:
This paper aims to describe the research protocol that will be used to determine the effectiveness of a health-social partnership intervention programme among community-dwelling older adults

DETAILED DESCRIPTION:
A staff of community center in service area who will not take part in the study will be involved in drawing a list of potential participants from the accessible population. Simple random sampling will be adopted to recruit participants. Those who meet the inclusion and exclusion criteria and agree to participate in the research study will be assigned to intervention group or customary care group according to the result of randomization.

Sample size calculation was based on power analysis. Power analysis adopts a hypothesis-testing method to determine sample size according to several parameters which include pre-specified significance level, desired power level and expected effect size. Assuming a two-tailed alpha of 0.05, a probability of 0.2 for beta error (80% power), and an effect size of 0.28 after calculating with respect to the same primary outcome measure (self-efficacy) from results of two previous researches which provide home visit and telephone follow up to older adults, 200 subjects per group are required. With reference to the 10% to 15% attrition reported in previous community-dwelling elderly program, assume there is a 20% drop out rate in this study, the total sample size needed is 240 subjects per group i.e. a total of 480 subjects.

In order to assure that the numbers of both groups are equal, a block randomization method will be used. Before randomization, a project team member who will not be involved in the subject recruitment and data collection will prepare a block randomization list with 240 sets of numbers which is either 0 (customary care group) or 1 (intervention group) by using a computer software Research Randomizer (http://www.randomizer.org/). These 240 sets of numbers will be printed out separately and sealed in each envelope. Another project team member, who successfully recruits a subject, will unfold an envelope by sequence after the enrolled participants finished all the baseline assessment and ready for interventions. The number written in the envelope will represent the group of that particular subject.

The group assignments will keep blinded to participants during the whole study period. However, the nurse case manager who will provide care to the participants will know the group allocation. Therefore, this study is a single-blinded design. In order to minimize bias, the nurse case manager will not participate in the data collection procedure.

Descriptive analysis will be calculated using mean and standard deviation for continuous variables, percentage and frequency for categorical variables, and median and quartile range when the continuous variables are not normally distributed. Independent t-tests, Mann-Whitney U test, chi-square test or Fisher's exact test will be used to compare any differences in socio-demographic data or outcome variables between groups. Significant results are indicated if p-value of all statistical analysis is less than 0.05 for two-tailed test. To determine the differences or changes between study group and control group (between group effects), within group effects (time), and the interaction effects (group x time), two way repeated measures Analysis of variances (ANOVA) or co-variances (ANCOVA) will be applied when assumptions for parametric test are fulfilled. When the data cannot fulfill the assumptions of parametric test, Mann-Whitney U test will be applied to compare the differences between groups at each time interval while Friedman test will be used to determine the time effects within each group.

The missing data in the present study will be handled by intention-to-treat (ITT) analysis. Sensitivity analysis will be adopted to compare the results using different missing data handling approach according to the Crochrane Handbook for Systematic Reviews of Interventions. Data will be computed and analyzed with the assistant of the Statistical package of Social Sciences (SPSS) version 21 software (SPSS Inc., Chicago).

All questionnaires for measuring the outcome variables in this study have been demonstrated good validity and reliability. Nurse case managers and social workers will be trained by the research team members in order to provide consistent interventions from various professionals in the health-social care team and ensure the quality of the program. The nurse case managers will be employed with a criterion of experienced community nursing background. The process of home visits and telephone conversation will be recorded for review and evaluation. The research team members and health-social care team members will have meeting regularly to discuss the cases so as to ensure the practice is aligning with the protocols. This randomized controlled study will also stringently follow the Consolidated Standards of Reporting Trials (CONSORT) statement.

ELIGIBILITY:
Inclusion Criteria:

* People aged 60 or above
* Living within the service area
* Cognitively competent with Chinese version Mini-Mental Status Examination (C-MMSE) with score ≥ 20 (Wong, et al., 2011)

Exclusion Criteria:

* Not communicable
* Bed bound
* Not reached by phone
* With psychiatric problems
* Already engaged in structured health or social programs
* Will not stay in Hong Kong for the current two months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will measure the community living older adults the change from baseline in self-efficacy belief in self-care management at home at 3-months and 6-months | pre-intervention, 3-month, 6-month
  All 10-item in the Chinese version are rated on a 4-point Likert scale ranging from 1= not at all true to 4= exactly true. Scores on the scale are summated and higher scores indicate greater self-efficacy.Measuring general self-efficacy can provide a way to evaluate the effectiveness of empowerment interventions.

SECONDARY OUTCOMES:
the change of medication adherence to chronic medications from baseline to 3-months and 6-months for community-living older adults | pre-intervention, 3-month, 6-month
  The outcome measure of medication adherence in this study is determined using 8-item Morisky Medication Adherence Scale (MMAS-8). This measure is designed to facilitate the recognition of barriers to and behaviors (either intentional or unintentional) associated with adherence to chronic medications such as anti-diabetic and anti-hypertensive drugs.
the change from baseline in physical activity level of community living older adults at 3-months and 6-months | pre-intervention, 3-month, 6-month
  physical activity level of the participants will be measured by the Physical Activity Level for the Elderly (PASE). PASE is a short and easily scored questionnaire that assesses the level of self-reported physical activity of people aged 65 years or older. It comprises 12-item measuring the frequency, duration, the energy spent and the amount of physical activities undertaken over the previous seven days.
the change from baseline in activity of daily living level at 3-months and 6-months | pre-intervention, 3-month, 6-month
  the Modified Barthel index will be used to measures a person's performance in 10 activities of daily living functions using a 5-point Likert scale from 1= total dependent to 5= fully independent. These 10 items are feeding, dressing, grooming, bathing, toileting, bed-chair transfer, bladder and bowel control, ambulation and stair climbing.
the change from baseline in Instrumental activity of daily living level at 3-months and 6-months | pre-intervention, 3-month, 6-month
  the Chinese version of The Lawton Instrumental Activities of daily living scale will be used in assessing the complex activities performance of older adults. It is a four-point scale with 9-items of activities which include use of telephone, transportation, shopping, meal preparation, housework, handyman work, laundry, medication management, and money management.
nutritional status of community-living older adults from pre-intervention to post intervention at 3-months and 6-months | pre-intervention, 3-month, 6-month
  The nutritional status of older adults will be measured by the short form of Mini Nutritional Assessment (MNA-SF). The tool comprises six questions which cover the areas of weight, appetite and activity.
the chnage of perception of quality of life from baseline to at 3-months and 6-months post-intervention | pre-intervention, 3-month, 6-month
  Quality of life of community-living older adults is measured by SF-12 questionnaires. This questionnaire is a generic measure, as opposed to one that targets a specific age and disease. It has shown useful in Chinese elderly patients.
the change of depression level of community living older adults from baseline to at 3-months and 6-months post-intervention | pre-intervention, 3-month, 6-month
  The Chinese version of Geriatric depression scale is used to assess the depressive symptoms of community-dwelling older people. The questionnaire consists of 15 questions which are used to explore the feelings of participants with the dichotomous answers.
change from baseline in life satisfaction of community living older adults at 3-months and 6-months | pre-intervention, 3-month, 6-month
  A five-point scale of Global item of life satisfaction is used to measure the Life satisfaction of participants. It has shown a high correlation with a multi-dimensional life satisfaction scale.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, Msc, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Salvation army, Kowloon, Hong Kong

REFERENCES:
- [Result] Wong GK, Lam SW, Wong A, Lai M, Siu D, Poon WS, Mok V. MoCA-assessed cognitive function and excellent outcome after aneurysmal subarachnoid hemorrhage at 1 year. Eur J Neurol. 2014 May;21(5):725-30. doi: 10.1111/ene.12363. Epub 2014 Jan 28. PMID 24471651
- [Result] Wong FK, Ho MM, Yeung S, Tam SK, Chow SK. Effects of a health-social partnership transitional program on hospital readmission: a randomized controlled trial. Soc Sci Med. 2011 Oct;73(7):960-9. doi: 10.1016/j.socscimed.2011.06.036. Epub 2011 Jul 22. PMID 21839564
- [Result] Wong FK, Chow SK, Chan TM, Tam SK. Comparison of effects between home visits with telephone calls and telephone calls only for transitional discharge support: a randomised controlled trial. Age Ageing. 2014 Jan;43(1):91-7. doi: 10.1093/ageing/aft123. Epub 2013 Aug 26. PMID 23978408
- [Result] Nicolaides-Bouman A, van Rossum E, Habets H, Kempen GI, Knipschild P. Home visiting programme for older people with health problems: process evaluation. J Adv Nurs. 2007 Jun;58(5):425-35. doi: 10.1111/j.1365-2648.2007.04235.x. Epub 2007 Apr 17. PMID 17442032
- [Result] Yoo H, Kim CJ, Jang Y, You MA. Self-efficacy associated with self-management behaviours and health status of South Koreans with chronic diseases. Int J Nurs Pract. 2011 Dec;17(6):599-606. doi: 10.1111/j.1440-172X.2011.01970.x. PMID 22103826